CLINICAL TRIAL: NCT06674512
Title: Evaluating the Effectiveness of Pharmaceutical Service for Inpatient with Drug-related Problems（INPATDRP）: a Randomized Controlled Trial
Brief Title: The Effectiveness of Pharmaceutical Service for INPATDRP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KY2024148
Record Dates: First submitted 2024-10-27; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Drug Related Problem
Keywords: Drug Related Problem; Inpatient; Clinical Pharmacist

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinical Pharmacist-led Pharmaceutical Services (Experimental): In addition to usual care services, the intervention group was provided with pharmaceutical care by a clinical pharmacist.
  Interventions: Behavioral: Clinical Pharmacist-led Pharmaceutical Services
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Clinical Pharmacist-led Pharmaceutical Services — Pharmacists developed an intervention plan to reduce DRPs and improve patients' quality of life by assessing patients' medication knowledge, drug-related problems, and adherence problems in the intervention group in the order of urgency, importance, and priority to be addressed. The plan included a list of patients' medication or lifestyle-related problems, a list of programs based on the assessed problems, and other information.
  Arms: Clinical Pharmacist-led Pharmaceutical Services

SUMMARY:
Medication risk is defined as the potential for loss or harm that may result from the use of medications during the course of treatment. Drug-related problems (DRPs) are defined as events or situations involving drug therapy that actually or potentially interfere with desired health outcomes. DRPs represent a significant aspect of medication risk in hospitalized patients, and the study and management of DRPs can effectively reduce the incidence of medication risk. DRPs are associated with both therapeutic efficacy and adverse drug events, and the timely identification and reduction of DRPs can enhance clinical efficacy and prevent the occurrence of adverse events.

DRPs pose a challenge to the clinician, and that may affect patient's clinical outcomes and may result in morbidity or mortality and increased health care costs. Health care costs may become a burden to the patient or may be to the government or to the third parties. Clinical Pharmacy is a discipline that promotes the quality use of medicines through evidence-based medicine and helps in identification and resolving DRPs. A clinical pharmacist through his/her clinical accuracy checking may identify DRPs and come out with suitable solutions to resolve the same.

Consequently, the aims of our study were to investigate the efficacy and safety effects of pharmacist-implemented drug-related problems (DRPs)-based interventions on patients' medication therapy.

DETAILED DESCRIPTION:
The study was conducted as a parallel randomized controlled study in a large general hospital in China.The study planned to enroll 220 inpatients aged 18 to 100. Subjects were randomly assigned to the intervention and control groups. Pharmacists managed patients' medications using a process for solving problems. This included:

1. Collecting information, assessing the patient's condition, and checking the medication plan.
2. Identifying and solving problems with medications.
3. Providing guidance on medications and creating personal medication lists.
4. Following up and reassessing. For patients in the intervention group, medication therapy management was done at the first visit. This included assessment, information collection, and possible interventions at the first visit and at the 1, 3, and 6 month follow-up visits. In the control group, patients were assessed at the first visit and at the 1, 3, and 6month follow-up visits. Information was collected, dosage and contraindications were explained, and necessary interventions were performed in the third month.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized patients;
2. Hospitalization duration >3 d;
3. Adult patients aged ≥18 years and ≤100 years (only adult patients aged 18 years or older were included in the medication management study because of the difference in study methodology between minor and adult patients);
4. Patients or close relatives gave informed consent and were willing to communicate with the clinical pharmacist and receive medication life education.

Exclusion Criteria:

1. Those who did not meet the inclusion criteria;
2. Patients who are in the acute phase of the disease requiring emergency medical consultation;
3. Those with any serious or life-threatening diseases (heart, lung, liver, kidney failure, hematologic diseases, malignant tumors, etc.);
4. Patients with psychiatric disorders, hearing impairments, intellectual disabilities, aphasia, etc. that make them unable to communicate or comply with the study protocol;
5. Any other reasons that the investigator believes may affect the efficacy and safety evaluation of this study other reasons not suitable for participation in this clinical trial (including, but not limited to, the investigator's judgment that the subject lives far away and is unable to follow up as scheduled).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of DRPs | One year from inclusion
  Number of drug related problems identified in inpatient
Change in DRPs | One year from inclusion
  Determination of drug-related problems (DRP) using Pharmaceutical Care Network Europe (PCNE) Version 9.1. The basic classification has 3 primary domains for problems, 9 primary domains for causes and 5 primary domains for Planned Interventions, 3 primary domains for level of acceptance (of interventions) and 4 primary domains for the Status of the problem.

SECONDARY OUTCOMES:
Medication Adherence | One year from inclusion
  The Morisky Adherence Scale was used, with scores less than 6 being low adherence, 6-7.75 being moderate adherence, and 8 being high adherence.
Patients' knowledge | One year from inclusion
  Using the medication knowledge evaluation tool, medication knowledge evaluation questionnaire with 7 questions,The patient scores 1 point if he/she knows the correct answer, 0 points if he/she does not know and -1 if the information given is incorrect. Score goes from -7 (patient who answers all questions incorrectly) to 7 (patient who answer all questions correctly) for each medication that the patient is taking. A score of 0 has no particular significance, apart from being in the middle of the two extremes.
Patient satisfaction in the experimental group | One year from inclusion
  Patient satisfaction in the intervention group was assessed using a patient satisfaction questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang Provincial, China

IPD SHARING:
Plan to Share IPD: No